CLINICAL TRIAL: NCT05150171
Title: Usability of an E-self-management Program for Treatment of Hand Osteoarthritis - the Happy Hands Pilot Study
Brief Title: Happy Hands E-self-management Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: The Norwegian Rheumatism Association (Other)
Responsible Party: Principal Investigator, Anne Therese Tveter, Senior researcher, Diakonhjemmet Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REK 249364
Record Dates: First submitted 2021-11-26; First posted 2021-12-08 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Hand Osteoarthritis

STUDY DESIGN:
Intervention Model Description: An e-self-management intervention consisting of videos informing patients with hand osteoarthritis about recommended treatment (information, hand exercises, use of assistive devices and orthoses, information about pharmacological and surgical treatment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- e-self-management intervention (Experimental): Patients will receive the HAPPY Hands e-self-management intervention delivered through a smartphone app.
  Interventions: Other: e-self-management intervention

INTERVENTIONS:
Other: e-self-management intervention — The app is developed based on a combination of behavioural change techniques informed by Social cognitive theory and the EULAR recommendations on management of hand osteoarthritis. The 12-week intervention consists of 25 short informational videos addressing the themes prioritized by the patient research partners. Additionally, the intervention includes a hand exercise program consisting of 8 videos providing instructions on warm up, exercises to improve mobility, strength and coordination, and a stretching exercise. The informational videos and exercise program are delivered in a progressive order across the 12 weeks. Encouragement and motivational messages are provided each week to enhance continued adherence to the intervention.

SUMMARY:
This pilot study will assess usability of a e-self-management program for patients with hand osteoarthritis through the Happy Hands app. People with hand osteoarthritis will be recruited for the study. The e-self-management intervention consists of informational videos and videos of hand exercises and has a duration of 12 weeks. Patient-reported outcomes and grip strength will be collected before and after the 12 week intervention period. Change in pain, stiffness, grip strength, disease activity and quality indicators will be assessed after 12 weeks.

DETAILED DESCRIPTION:
Patients diagnosed with hand osteoarthritis will be recuited from The Norwegian Rheumatism Association, Diakonhjemmet Hospital and Ankerløkka Legesenter (general practitioner). Patients will be summoned for an appointment at Diakonhjemmet or another suitable place for testing of grip strength and instructions on how to download the app. The e-self-management intervention is a 12 week intervention delivered through the Happy Hands app.

The app is developed based on a combination of behavioural change techniques informed by Social cognitive theory and the EULAR recommendations on management of hand OA. The 12-week intervention consists of 25 short informational videos addressing the themes prioritized by the patient research partners. These themes are further operationalized into the following categories: "Information on hand OA", "Hand exercises", "Use of assistive devices and orthoses", "Medication and surgical alternatives", and "Self-management of the disease". Additionally, the intervention includes a hand exercise program consisting of 8 videos providing instructions on warm up, exercises to improve mobility, strength and coordination, and a stretching exercise. The informational videos and exercise program are delivered in a progressive order across the 12 weeks. When downloading the app, participants are asked to specify when they plan to use the app (three days a week with time points). Thereafter, patients get a notification on their smartphone with that week's informational videos and hand exercises on the specified days.

After each exercise session patients are asked to rate their pain and stiffness, and these answers are put into graphs visualising the development over the 12-week intervention period. Each month, patients also answer questions about hand function, which they can use to self-monitor their development across the intervention period. Encouragement and motivational messages are provided each week to enhance continued adherence to the intervention. Additionally, at the end of each week the patients are asked questions related to the informational videos the paticipants have seen that week for the purpose of promoting self-efficacy.

The primary aim is to assess the change in quality indicators from baseline to 12 weeks follow-up. Secondary aims are to assess the change in pain, stiffness, activity performance and grip strength from baseline to follow-up, and to assess the use of and adherence to the content of the app.

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with hand osteoarthritis
* Possessing a smartphone

Exclusion Criteria:

* cognitive deficits
* are scheduled for hand surgery within the next 3 months
* if they do not talk or understand Norwegian,
* if they have uncontrolled serious comorbidities.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Most women
Enrollment: 72 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in quality indicators for hand osteoarthritis treatment | Baseline and 12 week follow-up
  Quality indicators based on the OA-QI questionnaire, adopted to fit the treatment recommendations of hand osteoarthritis. 16 questions answered with yes, no or not appriopriate/do not know. Measured as pass rate.

SECONDARY OUTCOMES:
Pain intensity | Baseline and 12 week follow-up
  Numeric rating scale (0-10), 0=no pain, 10= worst possible pain
Pain intensity | After each exercise session (3 times a week for 12 weeks)
  Numeric rating scale (0-10), 0=no pain, 10= worst possible pain
Stiffness | Baseline and 12 week follow-up
  Numeric rating scale (0-10),0=no stiffness, 10= worst possible stiffness
Stiffness | After each exercise session (3 times a week for 12 weeks)
  Numeric rating scale (0-10),0=no stiffness, 10= worst possible stiffness
Grip strength | Baseline and 12 week follow-up
  Measured with Jamar dynamometer (kg), mean of two measures for each hand
Measure of Activity performance (MAP-Hand) | Baseline, 4 weeks, 8 weeks, 12 weeks follow-up
  18 questions conserning activity performance of the hand (1=no problem, 4=cannot do the activity), mean score from 1-4.
Quality indicators for hand osteoarthritis treatment | Baseline and 12 week follow-up
  Quality indicators based on the OA-QI questionnaire, adopted to fit the treatment recommendations of hand osteoarthritis. 16 questions answered with yes, no or not appriopriate/do not know. Measured as pass rate.
eHealth literacy | Baseline
  Measured with the eHEALS questionnaire, Norwegian version. 8 questions conserning eHealth literacy (strongly disagree - strongly agree)
System Usability Scale (SUS) | 12 week follow-up
  Questionnaire assessing the usability of the Happy Hands app, 10 questions (strongly agree - strongly disagree), index from 0-100 where 100 is best score
Number of painful joints | Baseline
  Number of painful joints on left and right hand
Disease activity | Baseline, 4 weeks, 8 weeks, 12 weeks
  Numeric rating scale (0-10), 0=no disease activity; 10=high disease activity
Change in condition | 4 weeks, 8 weeks, 12 weeks
  Global rating of change scale, likert scale with 7 answer options from much better to much worse
Demographic variables | Baseline
  Age, gender, other painful joints, sivil status, education, previous hand surgery, comorbidities
Motivation for hand exercises | Baseline
  Numeric rating scale (0-10), 0=no motivation, 10=best motivation
Adherence to app content | 12 weeks
  Number of exercises performed (0-36 exercise sessions) and informational videos watched (0-12 weeks) during the intervention period. Collected from the app

CONTACTS AND LOCATIONS:
Overall Officials: Anne Therese Tveter, PhD, Principal Investigator — Diakonhjemmet Hospital
Locations (2):
- Norway (2):
  - Norwegian Rheumatology Association, Oslo, Please Select
  - Diakonhjemmet Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No
Individual participant data may be made available upon reasonable request to the principal investigator.

REFERENCES:
- [Derived] Tveter AT, Varsi C, Maarnes MK, Pedersen SJ, Christensen BS, Blanck TB, Nyheim SB, Pelle T, Kjeken I. Development of the Happy Hands Self-Management App for People with Hand Osteoarthritis: Feasibility Study. JMIR Form Res. 2024 Oct 29;8:e59016. doi: 10.2196/59016. PMID 39470716